CLINICAL TRIAL: NCT04536584
Title: Randomized Study Estimating the Impact of a Personalized and Remote Support Centered on Exercise and Physical Activity for Patients After Breast Cancer
Brief Title: Impact of Personalized and Remote Support Centered on Exercise and Physical Activity for Breast Cancer Patients
Acronym: eMOUVOIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Stimulab (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: eMOUVOIR-1901
Record Dates: First submitted 2019-06-05; First posted 2020-09-02 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Female
Keywords: Non metastatic breast cancer; Post breast cancer support; Physical activities
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: personalized coaching for physical activities (Experimental): This arm consists of providing patients with a personalized coaching focused on exercise and physical activity, with or without connected watch.
  Interventions: Other: Personalized Coaching (Arm A)
- Arm B: standard supportive approach (Active Comparator): The standard supportive approach will consist in recommendations made during visits with the oncologist. The delivery of post-treatment care by oncologists and their team systematically provide exercise advice patients including recommendations for strength training and aerobic activity.
  Interventions: Other: Standard supportive approach (Arm B)

INTERVENTIONS:
Other: Personalized Coaching (Arm A) — Patients will receive personalized physical activity coaching with an online digital platform to take online educational workshops and interact with other peers of the cohort with a online private forum. They will also have a connected watch that will measure several physical activity metrics.
  Arms: Arm A: personalized coaching for physical activities
Other: Standard supportive approach (Arm B) — Patients will receive the standard recommendations during their visits with the oncologist. The exercise recommendations include strength training and aerobic activities.
  Arms: Arm B: standard supportive approach

SUMMARY:
A study that evaluates the benefits of a personalized remote exercise and physical activity coaching compared with the standard supportive approach in terms of health-related quality of life at 12 months in breast cancer survivors treated in an adjuvant setting.

DETAILED DESCRIPTION:
A multicentric, phase III, randomized open-labelled study with two parallel groups which evaluates the benefits of a personalized remote exercise and physical activity coaching compared with the standard supportive approach in terms of health-related quality of life at 12 months in breast cancer survivors treated in an adjuvant setting.

Other objectives include:

* To evaluate the impact of the intervention on each dimension of the SF-36 at 12 months
* To evaluate the impact of the program on the health-related quality of life over time
* To evaluate the impact of the program on the practice of exercise and physical activity (EPA) at the recommended intensity (30min of moderate EPA, 5 days/week)
* To evaluate the impact of the program on:

  o fatigue, pain, depression, sleep, motivation for the practice, self-respect, biometric measures (including fat mass and lean mass), physical capacities, patient's satisfaction regarding the assigned program, occurrence of Adverse Events (AE) related to the treatment, professional life for patients who worked before the announcement of getting cancer and psychotropic and analgesic drug intake
* To evaluate the compliance to the program through the engagement score during the first 4 months (in the experimental group).
* To evaluate the impact of the program in terms of disease-free survival

Additional objectives on health economics include:

* To evaluate the efficiency of the personalized remote exercise and physical activity coaching compared with the standard supportive approach in BC survivors treated in an adjuvant setting.
* To characterize the health-state utility of BC survivors over time; assessing the association of change in health-utility with changes in other variables such as exercise and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18;
* Diagnosis of invasive non-metastatic breast cancer;
* 5 months (+/- 3 months) after the end of the treatment by surgery and/or radiotherapy and/or chemotherapy and/or other "short-term" systemic treatment : immunotherapy, PARP inhibitor, trastuzumab or TDM1 ; the continuation of hormonotherapy (more or less associated with an anti-CDK4/6), trastuzumab or TDM1 is possible during the study period;
* SF-36 filled in completely
* Medical certificate for sports practice delivered by a healthcare professional or oncologist. Neither the previous sports practice, nor the motivation for the proposed program is necessary to participate in the program.
* Agreement for follow-ups during the study period lasting 12 months;
* Ability to understand, read and write French;
* Patient covered by the French "Social Security" regime;
* Signed informed consent for the participation in the study, including the randomization with a 50%/50% chance of being allocated to one or the other group.

Exclusion Criteria:

* Relapse of invasive breast cancer (loco-regional relapse, contralateral relapse)
* Inability to exercise because of a severe handicap or vulnerability. These contraindications are left to the discretion of the healthcare professional assessing capacity (ex : severe malnutrition, pregnancy …);
* Metastatic cancer;
* Expressed preference for one arm;
* Inability to comply with follow-up (4 and 12 months) of the trial (geographical, social, medical or psychological reasons);
* Person under guardianship or curatorship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 824 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Quality of Life (QoL): SF 36 PCS | 1 year from the inclusion
  This study will evaluate, in each randomized group, the difference between the baseline score and the 12-month score of summary score of this questionnaire: PCS (Physical Component Summary)
Quality of Life (QoL): SF 36 MCS | 1 year from the inclusion
  This study will evaluate, in each randomized group, the difference between the baseline score and the 12-month score of summary score of this questionnaire: MCS (Mental Component Summary)

SECONDARY OUTCOMES:
Success/Failure score | at 12 months after start of the program
  For each summary score (PCS and MCS) separately, the success or failure score will be calculated :
  * For patients with an intermediate or good QoL at baseline (summary score≥50), failure is defined as a score decrease ≥ 5 points whereas a stable measure (difference of less than 5 points) and improvement of ≥ 5 points will be classified as a success.
  * For patients with a relatively poor QoL at baseline (summary score <50), success is defined as a score increase of 5 points or more at 12 months. All other cases are classified as a failure.
Health Related Quality of Life (HRQoL) | at the baseline, 4 months, 8 months and 12 months.
  The HRQoL evaluated with the Short-Form-36 questionnaire. We chose the SF-36 generic questionnaire to assess HRQoL of these patients instead of a cancer-specific HRQoL questionnaire such as the EORTC QLQ-C30. In fact, the QLQ-C30 as well as majority of cancer-specific questionnaires is focused on symptoms and side effects such as nausea and vomiting, which are not relevant for cancer survivorship. Thus, patients will not concerned by these items. The creation of an EORTC cancer survivorship questionnaire is ongoing, but this questionnaire is not validated yet at the time of the start of this study. Thus, a generic questionnaire, the SF-36, was considered as more relevant and sensitive to change for these patients.
Practice of Exercise and Physical Activities (EPA) | at the baseline, 4 months, 8 months and 12 months.
  The EPA will be evaluated with the Global Physical Activity Questionnaire for the patient's subjective measure and with the connected watch in the experimental arm for the objective measure.
  The Global Physical Activity Questionnaire is an instrument to assess physical activity. It was developed under the auspices of the WHO in 2002. GPAQ comprises 19 questions grouped to capture physical activity undertaken in different behavioral domains, these are work, transport and discretionary (also known as leisure or recreation). Within the work and discretionary domains, questions assess the frequency and duration of 2 differents categories of activity defined by the energy requirement or intensity. In the transport domain, the frequency and duration of all walking and cycling is captured but no attempt is made to differentiate between these activities. One additional item collected time spent in sedentary activities.
Fatigue | at the baseline, and 12 months.
  Will be evaluated with the Brief Fatigue Inventory auto-questionnaire The Brief Fatigue Inventory (BFI) is a questionnaire uses an 11-point scale (0 to 10) to measure the specific symptom of cancer-related fatigue in a single dimension. Nine items ask patients to rate the severity of their fatigue at its "worst," "usual," and "now" during the past 24 hours, with 0 = "no fatigue" and 10 = "fatigue". Cut points for fatigue severity are defined in two categories: a "fatigue worst" rating of 7 or greater indicates "severe" and 0 to 6 indicates "non-severe." Six additional items describe how much fatigue has interfered with different aspects of the patient's life during the past 24 hours. These items include general activity, mood, walking ability, normal work (includes both work outside the home and housework), relationships with other people, and enjoyment life.
Pain level | at the baseline, and 12 months.
  Will be evaluated with the Brief Pain Inventory-SF (Brief Pain Inventory-short form) auto-questionnaire The Brief Pain Inventory - Short Form (BPI-sf) is used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. It is a 9 item self-administered questionnaire. The patient is asked to rate their worst, least, average, and current pain intensity, list current treatments and their perceived effectiveness, and rate the degree that pain interferes with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life on a 10 point scale.
Depression | at the baseline, and 12 months.
  Will be evaluated with the Hospital Anxiety and Depression Scale auto-questionnaire The Hospital Anxiety and Depression Scale (HADS) is a self-administrated questionnaire to detect anxiety and depressive disorders, validated in French with a general population and suffering from cancer. It has 14 items with 4 answers proposed and each correspond to a score between 0 to 3. Seven questions relate to anxiety and seven others to depressive dimension, thus allowing two scores to be obtained (maximum score of each score = 21). For subscales, a score of 0 to 7 is an absence of disorders (anxiety or depressive, depending on the subscale), 8 to 10 to a suspected disorder and 11 to 21 to a proven disorder.
Sleep | at the baseline, and 12 months.
  Sleep will be evaluated in both arms using the Pittsburgh Sleep ≥Index (PSQI). In the experimental group, the number of hours of light and deep sleep will also be collected (connected watch).
  The Pittsburgh Sleep Quality Index (PSQI) is designed to measure sleep quality over a onemonth interval. It includes 19 self-rated questions that generate seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Component scores (range 0 to 3) are summed to provide a global sleep quality score (range 0 to 21); a score greater than five indicates poor sleep quality.
Biometric measures (impedance) | at the baseline, 4 months, 8 months and 12 months.
  Will be evaluated with the weight, BMI, fat mass, lean mass, waist size and hip size.
  These multiple measurements will be aggregated to arrive at one reported value, for exemple BMI.
Physical capacities | at the baseline, 4 months, 8 months and 12 months.
  Will be evaluated through differents physical exercices, for exemple:
  * Chair test (resistance test of lower limbs)
  * Weight test (resistance test of upper limbs)
  * Hand grip test (gripping force)
  * Goniometer test (flexibility of upper limbs)
  * Test of unipodal support (balance)
  * 6-min walking test
  * Heart rate by telemetry (Beating per minute - cardiac rhythm)
  * Borg Rating of Perceived Exertion Scale And these multiple measurements will be aggregated to arrive at one reported value.
Adverse Events | at the baseline, 4 months, 8 months and 12 months.
  Adverse Events graded according to NCI-CTC-AE v5, considering all types of AE, related to the evaluated program or to concomitant/previous anti-cancer treatments
Professional activity status | at the baseline, 4 months, 8 months and 12 months.
  Professional activity status before diagnosis and after anti-cancer treatment (temporary interruption, partial time work…).
  At baseline and during the follow-up, record the professional staut of the patients to provide the statistical trend regarding the professional activities.
Drug intake | at the baseline, 4 months, 8 months and 12 months.
  Will be evaluated with the frequency of psychotropic (including hypnotic) and analgesic intake
Disease-free survival | at the baseline, 4 months, 8 months and 12 months.
  Disease-free survival defined as the time between randomization and relapse or death from any cause.
Health states descriptive system | at the baseline, 4 months, 8 months and 12 months.
  Using EQ-5D and EQ VAS (study entry, M4, M8 and M12) and direct medical costs from inclusion up the M12.
  The descriptive system comprises five dimensions. Each dimension has five levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The respondent is asked to indicate her health state by ticking in the box against the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number expressing the level selected for that dimension. The digits for five dimensions can be combined in a 5-digit number describing the respondent's health state (for instance, " 11111 " corresponding to the perfect health).
  The EQ VAS records the respondent's self-rated health on a 20 cm vertical (graduate 0 to 100), visual analogue scale with endpoints labeled 'the best health you can imagine' and 'the worst health you can imagine'.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence VANLEMMENS, MD, Principal Investigator — Centre Oscar Lambret
Locations (22):
- France (22):
  - Centre Léon Bérard, Lyon, Auvergne-Rhône-Alpes
  - Groupe Hospitalier Bretagne Sud, Lorient, Brittany Region
  - CARIO Hôpital Privé des Côtes d'Armor, Plérin, Brittany Region
  - Centre Eugène marquis, Rennes, Brittany Region
  - Centre d'oncologie et radiothérapie Saint-Jean, Saint-Doulchard, Centre-Val de Loire
  - Sainte Catherine Institut du Cancer Avignon Provence, Avignon, France
  - Centre Marie Curie, Arras, Hauts-de-France
  - Centre Pierre Curie, Beuvry, Hauts-de-France
  - CH de Boulogne-sur-Mer, Boulogne-sur-Mer, Hauts-de-France
  - Centre de radiothérapie Amethyst, Compiègne, Hauts-de-France
  - Institut André Dutreix, Dunkirk, Hauts-de-France
  - Centre Oscar Lambret, Lille, Hauts-de-France
  - Centre Gray-Amethyst Radiothérapie, Maubeuge, Hauts-de-France
  - CH de Roubaix, Roubaix, Hauts-de-France
  - Centre Joliot Curie, Saint-Martin-Boulogne, Hauts-de-France
  - Centre de cancérologie Les Dentellières, Valenciennes, Hauts-de-France
  - CH de Valenciennes, Valenciennes, Hauts-de-France
  - Centre Hospitalier Eure-Seine - Hôpital d'Evreux, Évreux, Normandy
  - Institut Bergonié, Bordeaux, Nouvelle-Aquitaine
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux, Nouvelle-Aquitaine
  - Hôpital Privé du Confluent, Nantes, Pays de la Loire Region
  - Institut Gustave Roussy, Villejuif, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided